CLINICAL TRIAL: NCT04817046
Title: Detection of Early-stage Lung Cancer Based on Liquid Biopsy of Peripheral Blood: a Prospective Study
Brief Title: Assessment of Early-detection Based on Liquid Biopsy in Lung Cancer (ASCEND-LUNG)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Professor, Peking University People's Hospital
Other Study IDs: PTHO2101
Record Dates: First submitted 2021-03-10; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer
Keywords: Liquid Biopsy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and peripheral blood will be collected. Tissue DNA and cell-free DNA will be extracted for genetic analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a lung cancer diagnosis tool using a multi-omics approach based on liquid biopsy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a screening process to determine eligibility of study entry. Peripheral blood, tissue sample and imaging examinations of eligible patients will be collected for further analysis. Data collected will be used to develop a multi-omics lung cancer diagnosis model.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female, age equal to or greater than 40 years old and less than 75 years old
* Blood sample was collected before surgery for the detection of cfDNA methylation and other biomarkers
* Lung cancer patients diagnosed for the first time within 42 days before blood sampling without any anti-tumor treatment; or patients who are highly suspected of lung cancer through imaging evaluation or other routine clinical diagnosis and confirmed by tissue biopsy or surgical specimens within 42 days after blood sampling
* The subject has not received any local or systemic anti-tumor therapy before blood collection, including (not limited to) any surgery, local or systemic radiotherapy and chemotherapy, targeted therapy (including anti-angiogenesis), immunotherapy, cancer vaccines and hormone therapy, etc.

Exclusion Criteria:

* Unable to obtain sufficient and qualified blood samples
* Female subjects who are pregnant or breastfeeding
* Patients who have received organ transplantation or non-autologous bone marrow or stem cell transplantation
* Patients who have received blood transfusion within 7 days before blood sampling
* Patients who have received anti-infection treatment within 14 days before blood collection
* Patients who have receiving anti-tumor drugs for other diseases within 30 days before blood collection, such as methotrexate, cyclophosphamide, mercaptopurine, chlorambucil, tamoxifen, etc.
* Patients who suffered from other malignant tumors or multiple primary tumors at the same time
* Pathological confirmed benign lesions by tissue biopsy or surgery
* Insufficient sample for a confirmed pathological diagnosis
* Lung cancer patients with ground glass nodules on CT imaging.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed lung cancer patients between 40-75 years old, with solid nodule on CT imaging.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Estimated)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the multi-omics early-stage lung cancer diagnosis model | through study completion, an average of 1.5 year
  Sensitivity and specificity of the multi-omics early-stage lung cancer diagnosis model

SECONDARY OUTCOMES:
Accuracy of diagnostic models established separately from multi-omics data | through study completion, an average of 1.5 year
  Sensitivity and specificity models established separately from multi-omics data
Relationship between multi-omics data | through study completion, an average of 1.5 year
  Explore the relationship of features extracted from multi-omics data

CONTACTS AND LOCATIONS:
Overall Officials: Fan Yang, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jin Y, Mu W, Shi Y, Qi Q, Wang W, He Y, Sun X, Yang B, Cui P, Li C, Liu F, Liu Y, Wang G, Zhao J, Zhang Y, Zhang S, Cao C, Sun C, Hong N, Cai S, Tian J, Yang F, Chen K. Development and validation of an integrated system for lung cancer screening and post-screening pulmonary nodules management: a proof-of-concept study (ASCEND-LUNG). EClinicalMedicine. 2024 Aug 3;75:102769. doi: 10.1016/j.eclinm.2024.102769. eCollection 2024 Sep. PMID 39165498